CLINICAL TRIAL: NCT00431834
Title: Medtronic Concomitant Utilization of Radio Frequency Energy for Atrial Fibrillation (CURE-AF)/Permanent Study
Brief Title: Concomitant Utilization of Radio Frequency Energy for Atrial Fibrillation (CURE-AF) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURE-AF/Permanent
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-08

CONDITIONS: Atrial Fibrillation
Keywords: Permanent Atrial Fibrillation Surgical RF Ablation; Permanent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardioblate System Surgical Ablation System — This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.
Procedure: Surgical RF Ablation — This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.

SUMMARY:
This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with atrial fibrillation (AF) requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass graft (CABG) procedures. The study objectives are to demonstrate that the Medtronic Cardioblate Surgical Ablation System can safely and effectively treat permanent AF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a documented history of permanent AF (cardioversion failure) as defined by the ACC/AHA/ESC Guidelines.
2. Concomitant indication (other than AF) for open-heart surgery for one or more of the following:

   * Mitral valve repair or replacement
   * Aortic valve repair or replacement
   * Tricuspid valve repair or replacement
   * Atrial septal defect (ASD) repair
   * Patent foramen ovale (PFO) closure
   * Coronary artery bypass procedures
3. Greater than or equal to 18 years of age
4. Able and willing to comply with study requirements by signing a consent form
5. Must be able to take the anticoagulant warfarin (Coumadin)

Exclusion Criteria:

1. Wolff-Parkinson-White syndrome
2. NYHA Class = IV
3. Left ventricular ejection fraction ≤ 30%
4. Need for emergent cardiac surgery (i.e. cardiogenic shock)
5. Previous ablation for atrial fibrillation, AV-nodal ablation, or surgical Maze procedure
6. Contraindication for anticoagulation therapy
7. Left atrial diameter > 7.0 cm
8. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
9. Renal failure requiring dialysis or hepatic failure
10. Life expectancy of less than one year
11. Pregnancy or desire to be pregnant within 12 months of the study treatment.
12. Current diagnosis of active systemic infection
13. Documented MI 6 weeks prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thoralf Sundt, MD, Principal Investigator — The Mayo Clinic- Rochester
Locations (15):
- United States (15):
  - Southwest Heart and Lung, Phoenix, Arizona
  - East Bay Cardiovascular & Thoracic Associates, Concord, California
  - University of Southern California, Los Angeles, California
  - Eisenhower Medical Center, Palm Springs, California
  - Cardiac Surgical Associates of Florida, St. Petersburg, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Mayo/St. Mary's Hospital, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Lenox Hill Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Inova Fairfax, Falls Church, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Damiano RJ Jr, Badhwar V, Acker MA, Veeragandham RS, Kress DC, Robertson JO, Sundt TM. The CURE-AF trial: a prospective, multicenter trial of irrigated radiofrequency ablation for the treatment of persistent atrial fibrillation during concomitant cardiac surgery. Heart Rhythm. 2014 Jan;11(1):39-45. doi: 10.1016/j.hrthm.2013.10.004. Epub 2013 Oct 31. PMID 24184028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 91 subjects were consented to the study, of which 75 subjects received study treatment at 14 of the 15 investigational centers in the United States. The first subject was enrolled on May 22, 2007 and last patient enrolled on February 19, 2010.
Pre-assignment Details: No additional wash out, run-in, or transition was utilized during this study.
Groups:
- Cardioblate Surgical Ablation System: 75 subjects were enrolled and treated. 62 subjects completed the study through 6 month follow-up. 3 subjects died, 7 subjects withdrew from the study, 2 subjects missed the endpoint visit, and 1 subject was lost to follow-up.
Period: Overall Study
Arm/Group | Cardioblate Surgical Ablation System
Started | 75
Completed | 62
Not Completed | 13
Not completed — Withdrawal by Subject | 7
Not completed — Death | 3
Not completed — Missed Endpoint Visit | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Cohort: All subjects enrolled and treated with the Cardioblate Surgical Ablation System
Arm/Group | Entire Cohort
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 70.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: The Percent of Patients Off Class I and/or III Antiarrhythmic Drugs and Out of Atrial Fibrillation as Determined by 24 Hour Holter Recording Conducted at 6 Months Postoperatively.
Description: Subject's heart rhythm was evaulated by wearing a Holter Monitor for 24 hours.
Time Frame: 6 months
Population: 75 subjects were enrolled. 14 subjects had no holter analysis performed- 1 LTFU, 3 died,7 withdrew participation, 3 subjects without analyzable holter data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cardioblate Surgical Ablation System: All subjects enrolled who completed a Holter assessment at 6 month follow-up.
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 61
percentage of participants | 37.7 [25.3 to 50.1]
Statistical Analysis 1: Comparison: Cardioblate Surgical Ablation System; The specific test hypothesis is as follows: H0: ptest ≤ 22.1% Ha: ptest > 22.1%; Test type: Superiority or Other; p < 0.0041, Fisher Exact — The percent of patients off Class I and III AADs and successfully converted out of AF following treatment (ptest) will exceed the percenter of patients off Class I and III AADs and convereted out of AF, as reported in literature (pcontrol=22.1%); binomial proportions = 37.7, 97.5% CI 1-sided [lower limit 25.6]

2. Secondary Outcome: Efficacy Endpoints: The Percent of Patients Out of AF, Regardless of Antiarrhythmic Drug Status, as Determined by a 24 Hour Holter Recording at 6 Months
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Cardioblate Surgical Ablation System: All subjects enrolled who completed 6 month follow-up and had a 24-hour Holter assessment.
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 61
percentage of subjects | 63.9

3. Secondary Outcome: Safety Endpoints: Composite 6-month Major Adverse Event Rate, Post-procedure
Description: Major Adverse Events included: mediastinitis, death, myocardial infarction, stroke, transient ischemic attacks (TIA), pulmonary embolism, peripheral arterial embolism, and esophageal injury.
Time Frame: 6 months
Population: All subjects who were enrolled and were treated with the Cardioblate surgical ablation system with at least 6-month post-operative follow-up or an MAE prior to the end of the 6th month window were included in the analysis.
Measure: Number; unit: percentage of subjects
Groups:
- Cardioblate Surgical Ablation System: All subjects who were enrolled and were treated with the Cardioblate surgical ablation system with at least 6-month post-operative follow-up or an MAE prior to the end of the 6th month window were included in the analysis.
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 69
percentage of subjects | 8.7

4. Primary Outcome: Safety Endpoint: Composite Acute Major Adverse Event Rate, Within 30 Days Post-procedure or Hospital Discharge
Description: as for outcome 3
Time Frame: 30 days post procedure or hospital discharge
Population: Entire study population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 75
Percentage of subjects | 5.3 [0 to 11.1]
Statistical Analysis 1: Comparison: Cardioblate Surgical Ablation System; The specific test hypothesis is as follows: H0: p ≥ 23.6% Ha: p < 23.6%; Test type: Superiority or Other; p < 0.0001, Fisher Exact — The percent of subjects following treatment, p, who experience any of the MAEs during the first 30 days following surgery, or hospital discharge, whichever is longer will be less than 23.6%; binomial proportions = 5.3, 97.5% CI 1-sided [upper limit 13.1]

ADVERSE EVENTS:
Time Frame: Adverse events reported from treatment through 6 month follow-up.
Description: This study was overseen by a Data Safety Monitoring Board (DSMB) and a Clinical Events Committee (CEC). The DSMB made reviewed the data and recommendations regarding any safety concerns and also assessed the data from a risk/benefit perspective. The CEC reviewed and adjudicated MAEs and serious adverse events (SAEs)
Groups:
- Study Completion Cohort: 75 subjects were enrolled and treated. 62 subjects completed the study through 6 month follow-up. 4 subjects died, 8 subjects withdrew from the study, and 1 subject was lost to follow-up.
Arm/Group | Study Completion Cohort
Serious Adverse Events (participants affected / at risk) | 46/75
Other Adverse Events (participants affected / at risk) | 62/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Completion Cohort (N=75)
Anemia (Blood and lymphatic system disorders) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 3 (3)
Hemmorrhage (Blood and lymphatic system disorders) | 3 (4)
Infection/Sepsis (Blood and lymphatic system disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrioventricular Third Degree AV Heart Block (Cardiac disorders) | 6 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Insufficiency/Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Renal Insufficiency/Failure: Dialysis Required (Renal and urinary disorders) | 3 (3)
Renal Insufficiency/Failure: No Dialysis Required (Renal and urinary disorders) | 2 (2)
Respirator Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rhythms with potentially deleterious hemodynamic consequences requiring intervention (Cardiac disorders) | 8 (9)
Sick Sinus Syndrome (Cardiac disorders) | 3 (3)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Aystole (Cardiac disorders) | 2 (2)
Cerebellar Hemorrhage (Nervous system disorders) | 1 (1)
Hematoma- rt psoas muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Entrapped SWAN-GANZ Catheter (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Damaged PPM Lead (Cardiac disorders) | 1 (1)
Worstening Heart Failure (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Ventricular Septal Defect (Cardiac disorders) | 1 (1)
Ventricular Tachycardia/Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Femoral Atery Psuedoaneurysm (Vascular disorders) | 1 (1)
Increased Blood Pressure (Vascular disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Failure to Thrive (Gastrointestinal disorders) | 1 (1)
Post-op ileus/small bowel obstruction abdominal hernia repair (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Completion Cohort (N=75)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Congestive Heart Failure (Cardiac disorders) | 4 (4)
Infection/Sepsis (Infections and infestations) | 4 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 23 (23)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Renal Insufficiency/Failure: No Dialysis Required (Renal and urinary disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
* Slow/delayed enrollment
* Medical management of subjects by non-investigators leading to medication washout protocol deviations
* Missing endpoint data (attrition) due to cohort demographics (old age, dementia, relocation, etc.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less